CLINICAL TRIAL: NCT02366585
Title: The Effect of Locally Delivered Ciclosporin as an Adjunct to Healing After Treatment of Periodontal Pockets
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PerioC Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERIOC_CTP001
Record Dates: First submitted 2015-02-12; First posted 2015-02-19 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment with Ciclosporin (Experimental): Treatment of two periodontal pockets with ciclosporin gel Non-treatment of two periodontal pockets in same patient as comparator
  Interventions: Drug: Ciclosporin

INTERVENTIONS:
Drug: Ciclosporin — Ciclosporin gel applied to two periodontal pockets

SUMMARY:
The main purpose of the trial is to investigate the effect of locally delivered ciclosporin as an adjunct to non-surgical mechanical debridement in the treatment of chronic periodontitis and to compare it to mechanical debridement alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good general health
* 2 pairs of contralateral interproximal periodontal sites with probing depths of ≥7mm in single-rooted teeth not associated with furcations or root furrows.The test sites should have a distance of at least two teeth to the control sites.
* Teeth selected should have a vital pulp as determined by thermal or electric stimulation

Exclusion Criteria:

* Patients already included in other clinical trials involving therapeutic intervention (either medical or dental)
* Periodontal treatment during the last 6 months
* Antibiotic treatment 6 months prior to the start of the trial
* Antibiotic prophylaxis required for dental treatment
* Patients with acute infectious lesions in the areas of intended treatment
* Regular anti-inflammatory medication
* Known history of ciclosporin allergy
* Ongoing medication that may affect the clinical features of periodontitis
* Patients who are smokers
* Patients that are immuno-compromized or on immunosuppressive medication
* Patients who are pregnant or lactating

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-03; Primary Completion 2016-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth (PPD) | 3 months
  Mean change in probing pocket depth (PPD) from baseline to 3-month examination
Bleeding on Probing (BoP) | 3 months
  Change in BoP (measured as present or absent) from baseline to 3-month examination

CONTACTS AND LOCATIONS:
Overall Officials: Per Ramberg, PhD, Principal Investigator — Göteborg University
Locations (1):
- The Sahlgrenska Academy, University of Gothenburg, Gothenburg, Sweden